CLINICAL TRIAL: NCT00563524
Title: AN ASCENDING MULTIPLE DOSE STUDY OF THE SAFETY, TOLERABILITY, PHARMACOKINETICS, PHARMACODYNAMICS, AND CLINICAL EFFICACY OF ILV-094 ADMINISTERED SUBCUTANEOUSLY OR INTRAVENOUSLY TO SUBJECTS WITH PSORIASIS
Brief Title: Study Evaluating The Safety And Tolerability Of ILV-094 In Subjects With Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3199K2-1105; B1981002 (Other: Alias Study Number); 2009-012554-20 (EudraCT Number)
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — fezakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Placebo Comparator)
  Interventions: Drug: ILV-094

INTERVENTIONS:
Drug: ILV-094 — SC and IV administration on days 1, 14, 28, and 42
  Other Names: placebo

SUMMARY:
The purpose of this study is to assess safety, and tolerability of multiple doses of ILV-094 administered to subjects with psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Men and Women of nonchildbearing potential 18 years or older.
* Physician Area and Severity Index (PASI) greater than 11.
* Physician Global Assessment (PGA) greater than 3.

Exclusion Criteria:

* Use of any investigational small -molecule drug within 30 days before the first dose of test article administration, and use of any investigational biologic agents within 5 half lives before study day 1, or 90 days for investigational biologics that may have a long clinical duration of effect.
* Live vaccines within 3 months before test article administration or during the study.
* Use of any biologic therapy within approximately 5 half-lives before test article administration. Approximate half-lives of biologic therapies approved for psoriasis are as follows: Enbrel, 5 days; Humira, 14 days; Remicade, 9 days; Amevive, 12 days; Raptiva, 6 days. It is recommended that Amevive be discontinued for at least 90 days because of its long clinical duration of action.
* Psoralen plus ultraviolet A radiation (PUVA) therapy within 4 weeks before study day 1.
* Ultraviolet B (UVB) therapy within 2 weeks before study day 1.
* Receipt of systemic psoriasis therapy (eg, oral retinoids, methotrexate, hydroxyurea, cyclosporine, or azathioprine) or systemic corticosteroids within 4 weeks before study day 1.
* Topical steroids, topical vitamin A or D analog preparations, or anthralin within 2 weeks before study day 1. (Exception: topical therapies, including steroids at no higher than mild strength [class 6 or 7 topical corticosteroids], are permitted on the scalp, axillae, face, and groin, but the dose of the medication must be kept stable throughout the trial.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-12-20 (Actual); Primary Completion 2010-06-14 (Actual); Study Completion 2010-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (15):
  - David Stoll, MD, Beverly Hills, California
  - Dermatology Research, Santa Monica, California
  - Miami Research Associates, South Miami, Florida
  - MRA Clinical Research, South Miami, Florida
  - Hudson Dermatology, Evansville, Indiana
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Dawes Fretzin Dermatology Group, Indianapolis, Indiana
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Central Dermatology, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Duke Clinical Reseach Unit, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Baylor Research Institute, Dallas, Texas
- Canada (6):
  - Stratical Medical, Edmonton, Alberta
  - University of Alberta, Hospital Site Clinical Sciences Building, Edmonton, Alberta
  - The Northern Alberta Clinical Trials and Research Centre (NACTRC), Edmonton, Alberta
  - Bio Pharma Services Inc, Toronto, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Innovaderm Recherches Inc, Montreal, Quebec
- Queen Mary Hospital, Hong Kong, Hong Kong
- South Africa (2):
  - FARMOVS Parexel (Pty) Ltd, Bloemfontein, Free State
  - Parexel George, George, Western Cape

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=3199K2-1105

RESULTS

PARTICIPANT FLOW:
Groups:
- ILV-094 100 mg + 50 mg Subcutaneous: Participants received ILV-094 subcutaneous injections at a loading dose of 100 milligram (mg) on Day 1 and then 50 mg maintenance dose on Day 14, 28 and 42. Participants were followed up to 18 weeks.
- ILV-094 200 mg + 100 mg Subcutaneous: Participants received ILV-094 subcutaneous injections at a loading dose of 200 mg on Day 1 and then 100 mg maintenance dose on Day 14, 28 and 42. Participants were followed up to 18 weeks.
- Placebo Subcutaneous: Participants received placebo matched to ILV-094 subcutaneous injections on Day 1, 14, 28 and 42. Participants were followed up to 18 weeks.
- ILV-094 300 mg + 150 mg Intravenous: Participants received ILV-094 intravenous injections at a loading dose of 300 mg on Day 1 and then 150 mg maintenance dose on Day 14, 28 and 42. Participants were followed up to 18 weeks.
- ILV-094 600 mg + 300 mg Intravenous: Participants received ILV-094 intravenous injections at a loading dose of 600 mg on Day 1 and then 300 mg maintenance dose on Day 14, 28 and 42. Participants were followed up to 18 weeks.
- Placebo Intravenous: Participants received placebo matched to ILV-094 intravenous injections on Day 1, 14, 28 and 42. Participants were followed up to 18 weeks.
Period: Overall Study
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | Placebo Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous | Placebo Intravenous
Started | 13 | 12 | 13 | 12 | 13 | 13
Completed | 11 | 9 | 10 | 12 | 11 | 12
Not Completed | 2 | 3 | 3 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 3 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all randomized participants who received at least 1 dose of study medication.
Groups:
- ILV-094 100 mg + 50 mg Subcutaneous: Participants received ILV-094 subcutaneous injections at a loading dose of 100 mg on Day 1 and then 50 mg maintenance dose on Day 14, 28 and 42. Participants were followed up to 18 weeks.
- Total: Total of all reporting groups
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | Placebo Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous | Placebo Intravenous | Total
Number analyzed (Participants) | 13 | 12 | 13 | 12 | 13 | 13 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.54 (12.73) | 45.92 (10.15) | 44.46 (14.66) | 48.42 (14.02) | 47.69 (8.49) | 42.00 (15.55) | 44.43 (12.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 2 | 2 | 2 | 9
  Male | 13 | 11 | 11 | 10 | 11 | 11 | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) And Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; Initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug to the end of study (Day 126), that were absent before treatment or that worsened relative to pre-treatment state. AEs include both SAEs and all non-SAEs.
Time Frame: Day 1 up to Day 126
Population: Safety analysis population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | Placebo Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous | Placebo Intravenous
Number analyzed (Participants) | 13 | 12 | 13 | 12 | 13 | 13
Participants
  AEs | 3 | 9 | 7 | 11 | 9 | 9
  SAEs | 0 | 0 | 0 | 0 | 2 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Parameters
Description: Clinically significant ECG findings included: heart rate (HR): less than or equal to (<=) 45 beats per minute (bpm) or greater than or equal to (>=)120 bpm or decrease/increase of >=15 bpm from baseline value, PR interval: >=220 millisecond (msec) and change of >=20 msec from baseline value and; QRS interval >=120 msec; corrected QT (QTc) interval for men greater than (>) 450 msec, QTc interval for women >470 msec.
Time Frame: Day 1 up to Day 126
Population: Safety analysis population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | Placebo Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous | Placebo Intravenous
Number analyzed (Participants) | 13 | 12 | 13 | 12 | 13 | 13
Participants | 3 | 3 | 2 | 3 | 4 | 3

3. Primary Outcome: Number of Participants With Vital Sign Values of Potential Clinical Importance (PCI)
Description: Criteria for identifying vital sign values of PCI: heart rate: increase of >15 bpm from baseline value and >=120 bpm and decrease of >15 bpm from baseline value and <=45 bpm; Sitting and Supine systolic blood pressure (SBP): increase of >=20 millimeters of mercury (mm Hg) from baseline value and >=160 mm Hg and decrease of >=20 mm Hg from baseline value and <=90 mm Hg; Sitting and Supine diastolic blood pressure (DBP): increase of >=15 mm Hg from baseline value and >=100 mm Hg and decrease of >=15 mm Hg from baseline value and <=50 mm Hg; Respiratory rate: <10 or >25 breaths/minute; Weight: >=7 percent increase or decrease from baseline value; Oral temperature: <35 degree Celsius (C) or >38.3 degree C.
Time Frame: Day 1 up to Day 126
Population: Safety analysis population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | Placebo Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous | Placebo Intravenous
Number analyzed (Participants) | 13 | 12 | 13 | 12 | 13 | 13
Participants | 2 | 0 | 3 | 2 | 5 | 4

4. Primary Outcome: Number of Participants With Laboratory Test Values of Potential Clinical Importance
Description: Criteria:Hematocrit:5% decrease from baseline,Hemoglobin:decrease of >=20 gram per liter(g/L) from baseline,WBC: <3.0*10^9/L;neutrophils: <1.5*10^9/L,platelet count:<100*10^9/L,eosinophils: >0.5*10^9/L;prothrombin time,partial thromboplastin time: >1.5*Upper limit of normal(ULN);sodium,potassium: >5millimoles per liter(mmol/L)aboveULN/below lower limit of normal(LLN),creatinine: >1.36*ULN,urea: >1.5*ULN,glucose(fasting): >0.83mmol/L above ULN/below ULN,glucose (non-fasting): >5.0 mmol/L above ULN/>0.56 mmol/L below LLN,calcium:change of >=0.25 mmol/L from baseline,magnesium:change at >=0.21mmol/L from baseline value,phosphorus:>0.162 mmol/L above ULN/below LLN,total protein:change of >=20 g/L from baseline,albumin:change of >=10 g/L from baseline,uric acid:change of >0.119mmol/L from baseline,creatine kinase: >3*ULN,cholesterol: >7.77mmol/L,triglycerides:>3.39mmol/L;ALT,AST,total bilirubin: >2*ULN,alkaline phosphatase: >1.5*ULN,Gamma-glutamyl transferase,lactate dehydrogenase: >3*ULN.
Time Frame: Day 1 up to Day 126
Population: Safety analysis population included all randomized participants who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | Placebo Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous | Placebo Intravenous
Number analyzed (Participants) | 13 | 12 | 12 | 12 | 13 | 13
Participants | 10 | 10 | 7 | 10 | 7 | 7

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of ILV-094: Single Dose
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48, 96, 144, 192, 240, 312 hours post-dose on Day 1
Population: Pharmacokinetic (PK) analysis population included participants who received at least 1 dose of ILV-094 and had all available plasma concentrations and PK parameters.
Measure: Geometric Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous
Number analyzed (Participants) | 13 | 12 | 12 | 13
Microgram per milliliter | 6.292 (6.719) | 20.151 (32.716) | 79.475 (30.964) | 167.916 (32.488)

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of ILV-094: Multiple Dose
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 28, 96,144, 192, 240, 312, 480, 648, 816 hours post-dose on Day 14
Population: PK analysis population included participants who received at least 1 dose of ILV-094 and had all available plasma concentrations and PK parameters. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous
Number analyzed (Participants) | 11 | 10 | 12 | 11
Microgram per milliliter | 7.096 (5.138) | 19.222 (29.002) | 63.133 (21.736) | 113.523 (39.872)

7. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of ILV-094: Single Dose
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48, 96, 144, 192, 240, 312 hours post-dose on Day 1
Population: PK analysis population included participants who received at least 1 dose of ILV-094 and had all available plasma concentrations and PK parameters.
Measure: Median (Full Range); unit: Hour
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous
Number analyzed (Participants) | 13 | 12 | 12 | 13
Hour | 152.50 [48.0 to 263.9] | 107.77 [48.5 to 310.3] | 4.00 [1.0 to 314.1] | 3.00 [1.0 to 4.0]

8. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of ILV-094: Multiple Dose
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 28, 96,144, 192, 240, 312, 480, 648, 816 hours post-dose on Day 14
Population: as for outcome 6
Measure: Median (Full Range); unit: Hour
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous
Number analyzed (Participants) | 11 | 10 | 12 | 11
Hour | 48.07 [8.0 to 215.6] | 119.94 [47.2 to 263.8] | 2.00 [1.0 to 4.0] | 3.00 [0.0 to 24.0]

9. Secondary Outcome: Terminal-phase Disposition Rate Constant of ILV-094: Single Dose
Description: The terminal-phase disposition rate constant measured by a log-linear regression of the terminal mono exponential portion of the observed plasma concentrations, expressed in 1/day.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48, 96, 144, 192, 240, 312 hours post-dose on Day 1
Population: PK analysis set. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Standard Deviation); unit: One per day
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous
Number analyzed (Participants) | 13 | 12 | 8 | 12
One per day | NA (NA) — Data could not be calculated because values were below lower limit of quantification. | NA (NA) — Data could not be calculated because values were below lower limit of quantification. | 0.06623 (0.01438) | 0.08079 (0.01501)

10. Secondary Outcome: Terminal-phase Disposition Rate Constant of ILV-094: Multiple Dose
Description: as for outcome 9
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 28, 96,144, 192, 240, 312, 480, 648, 816 hours post-dose on Day 14
Population: as for outcome 9
Measure: Geometric Mean (Standard Deviation); unit: One per day
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous
Number analyzed (Participants) | 13 | 12 | 12 | 10
One per day | NA (NA) — Data could not be calculated because values were below lower limit of quantification. | NA (NA) — Data could not be calculated because values were below lower limit of quantification. | 0.04554 (0.00793) | 0.05302 (0.01163)

11. Secondary Outcome: Terminal Half-Life (t1/2) of ILV-094: Single Dose
Description: Plasma terminal half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48, 96, 144, 192, 240, 312 hours post-dose on Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous
Number analyzed (Participants) | 13 | 12 | 8 | 12
Days | NA (NA) — Data could not be calculated because values were below lower limit of quantification. | NA (NA) — Data could not be calculated because values were below lower limit of quantification. | 10.64 (1.99) | 8.69 (1.42)

12. Secondary Outcome: Terminal Half-Life (t1/2) of ILV-094: Multiple Dose
Description: Plasma terminal half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 28, 96,144, 192, 240, 312, 480, 648, 816 hours post-dose on Day 14
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous
Number analyzed (Participants) | 13 | 12 | 12 | 10
Days | NA (NA) — Data could not be calculated because values were below lower limit of quantification. | NA (NA) — Data could not be calculated because values were below lower limit of quantification. | 15.43 (2.68) | 13.45 (3.62)

13. Secondary Outcome: Area Under the Curve From Time Zero to The Time of Last Quantifiable Concentration (AUClast) of ILV-094: Single Dose
Description: AUClast is defined as area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 48, 96, 144, 192, 240, 312 hours post-dose on Day 1
Population: PK analysis population included participants who received at least 1 dose of ILV-094 with all available plasma concentrations and PK parameters.
Measure: Geometric Mean (Standard Deviation); unit: Hour*microgram per milliliter
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous
Number analyzed (Participants) | 13 | 12 | 12 | 13
Hour*microgram per milliliter | 1333 (1490) | 4212 (7783) | 8880 (2554) | 21358 (3696)

14. Secondary Outcome: Area Under the Curve From Time Zero to 312 Hours [AUC (0-312)] Postdose of ILV-094: Multiple Dose
Description: AUC (0-312) = Area under the plasma concentration time-curve from time zero (pre-dose) to 312 hours (0-312) postdose of ILV-094.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 28, 96,144, 192, 240, 312 hours post-dose
Population: PK analysis population included participants who received at least 1 dose of ILV-094 with all available plasma concentrations and PK parameters. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Standard Deviation); unit: Hour*microgram per milliliter
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous
Number analyzed (Participants) | 11 | 10 | 12 | 11
Hour*microgram per milliliter | 1532 (734) | 4241 (6434) | 9474 (3412) | 18352 (4810)

15. Secondary Outcome: Apparent Clearance of ILV-094: Multiple Dose
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after IV dose (apparent clearance) was influenced by the fraction of the dose absorbed.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 28, 96,144, 192, 240, 312, 480, 648, 816 hours post-dose on Day 14
Population: as for outcome 14
Measure: Geometric Mean (Standard Deviation); unit: Milliliter per hour
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous
Number analyzed (Participants) | 11 | 10 | 12 | 11
Milliliter per hour | 30.944 (20.160) | 22.536 (11.687) | 15.092 (4.832) | 15.586 (5.410)

16. Secondary Outcome: Apparent Volume of Distribution of ILV-094: Multiple Dose
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 28, 96,144, 192, 240, 312, 480, 648, 816 hours post-dose on Day 14
Population: as for outcome 9
Measure: Geometric Mean (Standard Deviation); unit: Milliliter
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous
Number analyzed (Participants) | 13 | 12 | 12 | 10
Milliliter | NA (NA) — Data could not be calculated because values were below lower limit of quantification. | NA (NA) — Data could not be calculated because values were below lower limit of quantification. | 7953 (1996) | 7174 (2283)

17. Secondary Outcome: Average Observed Plasma Concentration (Cavg) of ILV-094: Multiple Dose
Description: Cavg was the average plasma concentration of drug during the dosing interval.
Time Frame: Pre-dose, 1, 2, 3, 4, 8, 24, 28, 96,144, 192, 240, 312, 480, 648, 816 hours post-dose on Day 14
Population: as for outcome 14
Measure: Geometric Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous
Number analyzed (Participants) | 11 | 10 | 12 | 11
Microgram per milliliter | 4.809 (2.316) | 13.206 (20.301) | 29.580 (10.792) | 57.287 (14.946)

18. Secondary Outcome: Accumulation Ratio (Rac) of ILV-094
Description: Rac was estimated as: X*AUClast of Day 1 divided by AUC312 of Day 42, where X is the ratio of the maintenance dose to the loading dose of ILV-094, AUClast is defined as area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration and AUC-312 is the AUC from time 0 to 312 hours on Day 42.
Time Frame: Day 1: pre-dose, 1, 2, 3, 4, 8, 24, 48, 96, 144, 192, 240, 312 hours post-dose; Day 42: pre-dose, 1, 2, 3, 4, 8, 24, 28, 96,144, 192, 240, 312 hours post-dose
Population: as for outcome 14
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous
Number analyzed (Participants) | 11 | 10 | 12 | 11
Ratio | 2.739 (0.852) | 2.147 (1.283) | 2.134 (0.854) | 1.684 (0.375)

19. Secondary Outcome: Serum C-Reactive Protein (CRP) Levels
Description: CRP is an acute-phase protein which provides an objective criterion of inflammatory activity. Normal range of CRP is 0 milligram per deciliter (mg/dL) to 1 mg/dL. A decrease in the level of CRP indicates reduction in inflammation.
Time Frame: Day 1, 14, 28, 42, 56
Population: Pharmacodynamic (PD) analysis population included all randomized participants who received at least 1 dose of study medication and had all available PD. Here 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: Milligram per deciliter
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | Placebo Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous | Placebo Intravenous
Number analyzed (Participants) | 13 | 12 | 13 | 12 | 13 | 13
Milligram per deciliter
  Day 1: number analyzed (Participants) | 11 | 12 | 13 | 11 | 11 | 13
  Day 1 | 0.700 (1.075) | 1.943 (3.837) | 0.939 (2.017) | 0.446 (0.376) | 0.625 (0.672) | 1.142 (1.617)
  Day 14: number analyzed (Participants) | 11 | 12 | 12 | 12 | 13 | 12
  Day 14 | 0.742 (1.296) | 0.753 (0.666) | 0.972 (1.660) | 0.476 (0.399) | 0.587 (0.681) | 0.978 (1.401)
  Day 28: number analyzed (Participants) | 10 | 11 | 11 | 11 | 13 | 13
  Day 28 | 0.927 (1.147) | 1.001 (1.074) | 0.449 (0.481) | 0.435 (0.362) | 0.684 (0.494) | 0.870 (1.089)
  Day 42: number analyzed (Participants) | 11 | 10 | 11 | 11 | 12 | 12
  Day 42 | 0.703 (0.922) | 0.826 (1.048) | 0.424 (0.542) | 0.449 (0.493) | 0.691 (0.777) | 1.033 (1.447)
  Day 56: number analyzed (Participants) | 8 | 10 | 10 | 11 | 12 | 11
  Day 56 | 0.980 (1.372) | 1.158 (1.783) | 0.541 (0.474) | 0.393 (0.365) | 0.714 (1.121) | 1.100 (1.500)
Statistical Analysis 1: Comparison: ILV-094 100 mg + 50 mg Subcutaneous vs ILV-094 200 mg + 100 mg Subcutaneous vs ILV-094 300 mg + 150 mg Intravenous vs ILV-094 600 mg + 300 mg Intravenous; Baseline: Analysis of covariance (ANCOVA) with pre-dose as the baseline covariate and treatment as a factor was used for the analysis; Test type: Superiority or Other; p = 0.5237, ANCOVA
Statistical Analysis 2: Comparison: ILV-094 100 mg + 50 mg Subcutaneous vs ILV-094 200 mg + 100 mg Subcutaneous vs ILV-094 300 mg + 150 mg Intravenous vs ILV-094 600 mg + 300 mg Intravenous; Day 14: ANCOVA with pre-dose as the baseline covariate and treatment as a factor was used for the analysis; Test type: Superiority or Other; p = 0.8463, ANCOVA
Statistical Analysis 3: Comparison: ILV-094 100 mg + 50 mg Subcutaneous vs ILV-094 200 mg + 100 mg Subcutaneous vs ILV-094 300 mg + 150 mg Intravenous vs ILV-094 600 mg + 300 mg Intravenous; Day 28: ANCOVA with pre-dose as the baseline covariate and treatment as a factor was used for the analysis; Test type: Superiority or Other; p = 0.4596, ANCOVA
Statistical Analysis 4: Comparison: ILV-094 100 mg + 50 mg Subcutaneous vs ILV-094 200 mg + 100 mg Subcutaneous vs ILV-094 300 mg + 150 mg Intravenous vs ILV-094 600 mg + 300 mg Intravenous; Day 42: ANCOVA with pre-dose as the baseline covariate and treatment as a factor was used for the analysis; Test type: Superiority or Other; p = 0.6345, ANCOVA
Statistical Analysis 5: Comparison: ILV-094 100 mg + 50 mg Subcutaneous vs ILV-094 200 mg + 100 mg Subcutaneous vs ILV-094 300 mg + 150 mg Intravenous vs ILV-094 600 mg + 300 mg Intravenous; Day 56: ANCOVA with pre-dose as the baseline covariate and treatment as a factor was used for the analysis; Test type: Superiority or Other; p = 0.6235, ANCOVA

20. Secondary Outcome: Serum Interleukin-6 (IL-6) Levels
Time Frame: Day 1, 14, 28, 42, 56
Population: PD analysis population included all randomized participants who received at least 1 dose of study medication and had all available PD. Here 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: Picogram per milliliter
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | Placebo Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous | Placebo Intravenous
Number analyzed (Participants) | 13 | 12 | 13 | 12 | 13 | 13
Picogram per milliliter
  Day 1: number analyzed (Participants) | 8 | 12 | 11 | 8 | 8 | 10
  Day 1 | 3.14 (3.46) | 13.05 (22.01) | 4.93 (6.07) | 2.66 (1.65) | 2.46 (1.71) | 8.99 (18.53)
  Day 14: number analyzed (Participants) | 8 | 12 | 11 | 10 | 9 | 9
  Day 14 | 3.45 (3.80) | 8.05 (9.18) | 8.49 (15.92) | 2.08 (0.87) | 3.36 (3.05) | 8.16 (13.26)
  Day 28: number analyzed (Participants) | 7 | 11 | 10 | 9 | 11 | 7
  Day 28 | 4.17 (4.01) | 7.30 (6.76) | 3.41 (3.51) | 2.69 (1.87) | 3.51 (3.54) | 8.87 (12.65)
  Day 42: number analyzed (Participants) | 6 | 10 | 8 | 8 | 10 | 7
  Day 42 | 4.40 (4.93) | 8.34 (12.37) | 5.73 (6.45) | 2.09 (1.31) | 4.32 (4.19) | 10.41 (13.26)
  Day 56: number analyzed (Participants) | 6 | 10 | 9 | 7 | 7 | 9
  Day 56 | 2.43 (1.81) | 9.60 (11.80) | 4.90 (2.97) | 2.46 (1.47) | 6.19 (7.71) | 7.97 (12.87)
Statistical Analysis 1: Comparison: ILV-094 100 mg + 50 mg Subcutaneous vs ILV-094 200 mg + 100 mg Subcutaneous vs ILV-094 300 mg + 150 mg Intravenous vs ILV-094 600 mg + 300 mg Intravenous; Baseline: ANCOVA with pre-dose as the baseline covariate and treatment as a factor was used for the analysis; Test type: Superiority or Other; p = 0.3833, ANCOVA
Statistical Analysis 2: Comparison: ILV-094 100 mg + 50 mg Subcutaneous vs ILV-094 200 mg + 100 mg Subcutaneous vs ILV-094 300 mg + 150 mg Intravenous vs ILV-094 600 mg + 300 mg Intravenous; Day 14: ANCOVA with pre-dose as the baseline covariate and treatment as a factor was used for the analysis; Test type: Superiority or Other; p = 0.4909, ANCOVA
Statistical Analysis 3: Comparison: ILV-094 100 mg + 50 mg Subcutaneous vs ILV-094 200 mg + 100 mg Subcutaneous vs ILV-094 300 mg + 150 mg Intravenous vs ILV-094 600 mg + 300 mg Intravenous; Day 28: ANCOVA with pre-dose as the baseline covariate and treatment as a factor was used for the analysis; Test type: Superiority or Other; p = 0.2200, ANCOVA
Statistical Analysis 4: Comparison: ILV-094 100 mg + 50 mg Subcutaneous vs ILV-094 200 mg + 100 mg Subcutaneous vs ILV-094 300 mg + 150 mg Intravenous vs ILV-094 600 mg + 300 mg Intravenous; Day 42: ANCOVA with pre-dose as the baseline covariate and treatment as a factor was used for the analysis; Test type: Superiority or Other; p = 0.4183, ANCOVA
Statistical Analysis 5: Comparison: ILV-094 100 mg + 50 mg Subcutaneous vs ILV-094 200 mg + 100 mg Subcutaneous vs ILV-094 300 mg + 150 mg Intravenous vs ILV-094 600 mg + 300 mg Intravenous; Day 56: ANCOVA with pre-dose as the baseline covariate and treatment as a factor was used for the analysis; Test type: Superiority or Other; p = 0.4650, ANCOVA

21. Secondary Outcome: Serum Amyloid-A Levels
Time Frame: Day 1, 14, 28, 42, 56
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Picogram per milliliter
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | Placebo Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous | Placebo Intravenous
Number analyzed (Participants) | 13 | 12 | 13 | 12 | 13 | 13
Picogram per milliliter
  Day 1: number analyzed (Participants) | 13 | 11 | 13 | 12 | 11 | 12
  Day 1 | 26586201 (39787546) | 33048188 (45868899) | 22784245 (47173620) | 13112923 (13655594) | 32684269 (24358106) | 34103493 (33363700)
  Day 14: number analyzed (Participants) | 12 | 12 | 12 | 12 | 13 | 13
  Day 14 | 26708755 (51703518) | 37392805 (42940021) | 13930628 (9179161) | 15927358 (17100458) | 38017589 (27662906) | 55781761 (63622877)
  Day 28: number analyzed (Participants) | 12 | 11 | 11 | 12 | 12 | 13
  Day 28 | 16191087 (17818430) | 26521088 (22417132) | 11795968 (5741986) | 18546404 (26651017) | 40780444 (29197742) | 55618175 (47529302)
  Day 42: number analyzed (Participants) | 12 | 10 | 11 | 12 | 13 | 12
  Day 42 | 21215328 (28505898) | 19716955 (12180775) | 10203678 (8878853) | 19929741 (32444845) | 35032152 (27565726) | 60686782 (59133991)
  Day 56: number analyzed (Participants) | 9 | 9 | 11 | 12 | 13 | 11
  Day 56 | 9510659 (11632879) | 27246194 (23701114) | 17500314 (21390091) | 13943320 (14583899) | 35800358 (25684320) | 49462769 (58393285)
Statistical Analysis 1: Comparison: ILV-094 100 mg + 50 mg Subcutaneous vs ILV-094 200 mg + 100 mg Subcutaneous vs ILV-094 300 mg + 150 mg Intravenous vs ILV-094 600 mg + 300 mg Intravenous; Baseline: ANCOVA with pre-dose as the baseline covariate and treatment as a factor was used for the analysis; Test type: Superiority or Other; p = 0.7051, ANCOVA
Statistical Analysis 2: Comparison: ILV-094 100 mg + 50 mg Subcutaneous vs ILV-094 200 mg + 100 mg Subcutaneous vs ILV-094 300 mg + 150 mg Intravenous vs ILV-094 600 mg + 300 mg Intravenous; Day 14: ANCOVA with pre-dose as the baseline covariate and treatment as a factor was used for the analysis; Test type: Superiority or Other; p = 0.1072, ANCOVA
Statistical Analysis 3: Comparison: ILV-094 100 mg + 50 mg Subcutaneous vs ILV-094 200 mg + 100 mg Subcutaneous vs ILV-094 300 mg + 150 mg Intravenous vs ILV-094 600 mg + 300 mg Intravenous; Day 28: ANCOVA with pre-dose as the baseline covariate and treatment as a factor was used for the analysis; Test type: Superiority or Other; p = 0.0020, ANCOVA
Statistical Analysis 4: Comparison: ILV-094 100 mg + 50 mg Subcutaneous vs ILV-094 200 mg + 100 mg Subcutaneous vs ILV-094 300 mg + 150 mg Intravenous vs ILV-094 600 mg + 300 mg Intravenous; Day 42: ANCOVA with pre-dose as the baseline covariate and treatment as a factor was used for the analysis; Test type: Superiority or Other; p = 0.0079, ANCOVA
Statistical Analysis 5: Comparison: ILV-094 100 mg + 50 mg Subcutaneous vs ILV-094 200 mg + 100 mg Subcutaneous vs ILV-094 300 mg + 150 mg Intravenous vs ILV-094 600 mg + 300 mg Intravenous; Day 56: ANCOVA with pre-dose as the baseline covariate and treatment as a factor was used for the analysis; Test type: Superiority or Other; p = 0.0308, ANCOVA

22. Secondary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Scores at Week 2, 4, 6, 8 and 12
Description: PASI score is the combined assessment of lesion severity and area affected into single score range on a scale of 0 (no disease) to 72 (maximal disease), with higher scores indicating greater severity of psoriasis. Body divided into 4 sections (head and neck [h], arms [u], trunk [t], legs [l]); each area scored by itself and scores combined for final PASI score. For each section, percent body surface area (A) of skin involved was estimated: 0 (no involvement) to 6 (90-100 percent involvement), severity estimated by clinical signs: erythema (E), induration (I), scaling (S); 5 point scale: 0 (no involvement) to 4 (very marked involvement). Final PASI score = 0.1Ah (Eh + Ih + Sh) + 0.2Au (Eu + Iu + Su) + 0.3At (Et + It + St) + 0.4Al (El + Il + Sl), where head: 0.1; upper limbs: 0.2; trunk: 0.3; lower limbs: 0.4).
Time Frame: Baseline, Week 2, 4, 6, 8, 12
Population: PD analysis population included all randomized participants who received at least 1 dose of study medication and had all available PD and clinical disease evaluations. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows. Data were not collected at week 12 with subcutaneous administration.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | Placebo Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous | Placebo Intravenous
Number analyzed (Participants) | 13 | 12 | 13 | 12 | 13 | 13
Percent change
  Week 2 | 13.1 (17.3) | 13.5 (18.1) | 2.57 (9.29) | 14.0 (15.8) | 20.1 (14.9) | 11.3 (17.9)
  Week 4 | 11.4 (19.3) | 24.8 (34.0) | 6.36 (10.2) | 13.8 (16.7) | 32.6 (17.9) | 21.1 (20.3)
  Week 6 | 21.3 (21.6) | 19.3 (34.3) | 5.88 (16.0) | 30.3 (30.2) | 38.8 (21.4) | 25.8 (24.1)
  Week 8 | 27.3 (25.0) | 28.0 (34.6) | 8.71 (16.6) | 38.4 (38.6) | 39.4 (25.3) | 36.7 (39.1)
  Week 12: number analyzed (Participants) | 0 | 0 | 0 | 12 | 13 | 13
  Week 12 |  |  |  | 38.9 (41.5) | 38.3 (30.7) | 47.8 (38.4)

23. Secondary Outcome: Percent Change From Baseline in Target Lesion Score (TLS) at Week 2, 4, 6, 8 and 12
Description: TLS was based on the severity of 3 components: erythema, induration, and scaling. Severity of each component was evaluated on a 5-point scale as: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked, with higher scores reflected increased lesion severity. Scores of 3 components were summed to derive the total target lesion score, ranging from 0=none to 12=very marked, with higher scores reflected increased lesion severity.
Time Frame: Baseline, Week 2, 4, 6, 8, 12
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | Placebo Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous | Placebo Intravenous
Number analyzed (Participants) | 13 | 12 | 13 | 12 | 13 | 13
Percent change
  Week 2 | 1.38 (1.76) | 0.75 (1.21) | 1.00 (1.60) | 1.00 (1.21) | 1.69 (1.89) | 1.38 (1.66)
  Week 4 | 0.92 (1.56) | 1.58 (2.39) | 1.00 (1.48) | 1.83 (1.95) | 3.50 (2.24) | 2.38 (1.94)
  Week 6 | 1.83 (2.21) | 1.30 (2.26) | 1.18 (1.78) | 2.50 (2.28) | 3.75 (2.56) | 2.92 (2.15)
  Week 8 | 2.00 (2.83) | 1.80 (2.04) | 1.10 (1.20) | 3.08 (2.68) | 4.17 (2.52) | 2.83 (2.48)
  Week 12: number analyzed (Participants) | 0 | 0 | 0 | 12 | 13 | 13
  Week 12 |  |  |  | 3.27 (3.47) | 3.40 (2.17) | 3.75 (2.60)

24. Secondary Outcome: Percent Change From Baseline in Physician Global Assessment Score at Week 2, 4, 6, 8 and 12
Description: Physician global assessment of disease activity was measured on an 11-point scale, ranging from 0 = no disease activity to 10 = extreme disease activity, where higher scores indicating greater disease activity.
Time Frame: Baseline, Week 2, 4, 6, 8, 12
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | Placebo Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous | Placebo Intravenous
Number analyzed (Participants) | 13 | 12 | 13 | 12 | 13 | 13
Percent change
  Week 2 | 0.46 (0.78) | 0.33 (0.49) | 0.17 (0.39) | 0.55 (0.69) | 0.54 (0.52) | 0.23 (0.44)
  Week 4 | 0.25 (0.62) | 0.50 (0.67) | 0.18 (0.40) | 0.45 (0.52) | 1.08 (0.67) | 0.46 (0.66)
  Week 6 | 0.50 (0.67) | 0.50 (0.53) | 0.18 (0.40) | 0.73 (0.90) | 1.08 (0.90) | 0.75 (0.87)
  Week 8 | 0.82 (0.87) | 0.60 (0.52) | 0.20 (0.42) | 0.91 (0.94) | 1.25 (0.97) | 1.00 (0.95)
  Week 12: number analyzed (Participants) | 0 | 0 | 0 | 12 | 13 | 13
  Week 12 |  |  |  | 1.00 (0.82) | 1.10 (0.88) | 0.92 (0.90)

25. Other Pre Specified Outcome: Number of Participants With Positive Anti-Drug Antibodies Response
Description: Participants with their ADA titer levels >=6.23 were considered to be ADA positive. Participants with at least 1 positive ADA titer are reported.
Time Frame: Day 1 up to Day 126
Population: Safety analysis population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | Placebo Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous | Placebo Intravenous
Number analyzed (Participants) | 13 | 12 | 13 | 12 | 12 | 13
Participants | 0 | 0 | 0 | 3 | 0 | 1

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | ILV-094 100 mg + 50 mg Subcutaneous | ILV-094 200 mg + 100 mg Subcutaneous | Placebo Subcutaneous | ILV-094 300 mg + 150 mg Intravenous | ILV-094 600 mg + 300 mg Intravenous | Placebo Intravenous
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/13 | 0/12 | 2/13 | 0/13
Other Adverse Events (participants affected / at risk) | 3/13 | 9/12 | 7/13 | 11/12 | 9/13 | 9/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ILV-094 100 mg + 50 mg Subcutaneous (N=13) | ILV-094 200 mg + 100 mg Subcutaneous (N=12) | Placebo Subcutaneous (N=13) | ILV-094 300 mg + 150 mg Intravenous (N=12) | ILV-094 600 mg + 300 mg Intravenous (N=13) | Placebo Intravenous (N=13)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ILV-094 100 mg + 50 mg Subcutaneous (N=13) | ILV-094 200 mg + 100 mg Subcutaneous (N=12) | Placebo Subcutaneous (N=13) | ILV-094 300 mg + 150 mg Intravenous (N=12) | ILV-094 600 mg + 300 mg Intravenous (N=13) | Placebo Intravenous (N=13)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eyelid irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 0 | 1 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Arthroscopy (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 2 | 0 | 2 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Lymph node palpable (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary sediment present (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 2 | 2 | 2
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bromhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 3 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.